CLINICAL TRIAL: NCT02199483
Title: Metabolic and Neural Adaptations to Weight Loss, Plateau, and Regain
Status: Withdrawn | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 140154; 14-DK-0154
Record Dates: First submitted 2014-07-23; First posted 2014-07-24 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2017-06-29

CONDITIONS: Healthy Volunteers
Keywords: Energy Expenditure; Behavioral Weight Loss Treatment; Neurocognitive Function; Weight Loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Background:

- Many people can lose weight by changing their diet or exercise. However, most people eventually regain the weight over time. This weight regain may be related to changes in metabolism as well as changes in the brain caused by weight loss. Researchers want to learn more about these changes.

Objective:

- To see how weight loss and regain affects the body s metabolism and the brain of obese but healthy adults.

Eligibility:

- Obese but healthy adults age 18-55 who plan to participate in a weight loss program at one of several participating clinics or resorts.

Design:

* Participants will first be screened at home through questionnaires and telephone interviews.
* Participants will then be screened at the NIH with blood tests, medical history, physical exam, electrocardiograms, and questionnaires. They will have a mock magnetic resonance imaging (MRI) scan.
* At visit 1, participants will stay at the NIH and will:
* have MRI and PET brain scans.
* have body composition scans and measurements.
* give blood samples.
* eat a special diet.
* wear a physical activity monitor.
* provide a urine sample and body weight daily.
* drink a special type of water to measure calorie burn.
* wear a clear plastic hood over their head while lying down, to collect exhaled air.
* spend 24 hours in a room that measures oxygen and carbon dioxide.
* complete questionnaires and computer tasks.
* After visit 1, participants will give daily urine samples and weight and physical activity measurements from home. Then they will follow a lifestyle intervention for weight loss and give daily weight and activity measurements.
* Visits 2, 3, and 4 occur 1-26 months after the start of the weight loss program. Participants will repeat procedures from visit 1. Visits 1-4 last 4 days each.
* Researchers will track participants weight and physical activity for up to 26 months after visit 2.

DETAILED DESCRIPTION:
Lifestyle interventions can result in weight loss, but most people experience a plateau after 6-10 months when weight stabilizes and many subsequently regain weight over the subsequent months. This pattern of weight plateau and regain is typical and appears to be independent of the lifestyle intervention used. The apparent resistance to further weight loss in not well understood.

We recently demonstrated that participants engaged in an intensive intervention employing caloric restriction and vigorous exercise had a profound slowing of metabolism that was significantly greater than expected due to weight loss alone. This phenomenon is called metabolic adaptation and has also been observed following weight loss through caloric restriction without exercise and may persist long after weight loss has ceased. Metabolic adaptation has been hypothesized to limit weight loss and predispose individuals to weight regain, but this has yet to be demonstrated and the concept is controversial. In addition to the metabolic adaptations to weight loss, the brain also adapts in ways that enhance the activation of reward regions in response to palatable food cues and their receipt. In particular, the brain s dopamine circuitry is believed to be altered in obesity and it is presently unclear how this pathway responds to a weight loss intervention in humans.

The primary aims of this study are to investigate the metabolic and neural adaptations in 60 obese adult volunteers participating in lifestyle interventions resulting in weight loss through a structured meal replacement program or caloric restriction plus vigorous exercise. The secondary aim is to determine whether the magnitude of metabolic adaptation or the changes in the brain s reward circuitry or responsiveness to food cues are related to the ubiquitous weight loss plateau after 6-10 months or the rate of weight regain in the subsequent months.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age 18-55 years, male and female
* Recent weight stability (< plus and minus 2 % over past 1 month)
* Body mass index (BMI) greater than or equal to 30 kg/m2
* Able to complete daily bouts of moderate to vigorous exercise (when applicable)
* Written informed consent
* Have reserved a stay of at least 4 weeks at The Biggest Loser Resort or have enrolled in a structured meal replacement weight loss program at the Washington Center for Weight Management and Research, the National Center for Weight and Wellness, or the Johns Hopkins Weight Management Center.

EXCLUSION CRITERIA:

* Body weight > 400 lbs (weight limit of PET and MRI scanners)
* BMI < 30 kg/m2
* Less than 80% of maximum lifetime weight
* Hypertension if

  * (1) >160/100;
  * (2) 140/90 to 159/99 with evidence of target organ damage (e.g. elevated serum creatinine, proteinuria, abnormal EKG, retinopathy);
  * (3) >140/90 on antihypertensive medications.
* Evidence of metabolic or cardiovascular disease, or disease that may influence metabolism (e.g. cancer, thyroid disease)
* Past or present history of eating disorder (including binge eating) or psychiatric disease
* Taking any prescription medication or other drug that may influence metabolism (e.g. diet/weight-loss medication, asthma medication, psychiatric medications, corticosteroids, or other medications at the discretion of the PI and/or study team)
* Hematocrit < 34% (women only)
* Hematocrit < 40% (men only)
* Pregnancy, lactation (women only)
* Women who become pregnant during the two-year study period
* Recent participation in a regular exercise program (> 4h/week of vigorous activity)
* Previous bariatric surgery
* Caffeine consumption > 500 mg/day
* Regular use of alcohol (>2 drinks per day), tobacco (smoking or chewing) amphetamines, cocaine, heroin, or marijuana over past 6 months
* Volunteers with strict dietary concerns (e.g. vegetarian or kosher diet, multiple food allergies)
* Having metal implants incompatible with MRI (for example, pacemakers, metallic prostheses such as cochlear implants or heart valves, shrapnel fragments, etc.).
* Non-native English speakers
* Volunteers unwilling or unable to give informed consent

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-07-21; Primary Completion 2017-06-29 (Actual); Study Completion 2017-06-29 (Actual)

PRIMARY OUTCOMES:
To measure metabolic and neural adaptations after 4-12 weeks, 6-10 months, and 22-26 months following the start of a lifestyle intervention resulting in weight loss. | ongoing

SECONDARY OUTCOMES:
To determine whether the degree of metabolic or neural adaptation at 4-12 weeks is correlated with the weight plateau at 6-10 months or the rate of weight regain in the subsequent months. | ongoing
To investigate changes in circulating hormone and metabolites that correlate with metabolic and neural adaptations as well as changes in appetitive behaviors following a lifestyle intervention resulting in weight loss. | ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Hall, Ph.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)

REFERENCES:
- [Background] Franz MJ, VanWormer JJ, Crain AL, Boucher JL, Histon T, Caplan W, Bowman JD, Pronk NP. Weight-loss outcomes: a systematic review and meta-analysis of weight-loss clinical trials with a minimum 1-year follow-up. J Am Diet Assoc. 2007 Oct;107(10):1755-67. doi: 10.1016/j.jada.2007.07.017. PMID 17904936
- [Background] Arone LJ, Mackintosh R, Rosenbaum M, Leibel RL, Hirsch J. Autonomic nervous system activity in weight gain and weight loss. Am J Physiol. 1995 Jul;269(1 Pt 2):R222-5. doi: 10.1152/ajpregu.1995.269.1.R222. PMID 7631897
- [Background] Johannsen DL, Knuth ND, Huizenga R, Rood JC, Ravussin E, Hall KD. Metabolic slowing with massive weight loss despite preservation of fat-free mass. J Clin Endocrinol Metab. 2012 Jul;97(7):2489-96. doi: 10.1210/jc.2012-1444. Epub 2012 Apr 24. PMID 22535969